CLINICAL TRIAL: NCT02402400
Title: Sub Lingual Versus Traditional Oral Administration of Ticagrelor in Acute Coronary Syndrome
Brief Title: Sub Lingual Versus Traditional Oral Administration of Ticagrelor in Acute Coronary Syndrome/Non ST-elevation Myocardial Infarction - A Platelet Reactivity Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Elad Asher, MD, MHA, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-2028-15-SMC-EA-CTIL
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Acute Coronary Syndromes; Non ST Elevation Myocardial Infarction
Keywords: NSTEMI
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Ticagrelor (Active Comparator)
  Interventions: Drug: Sub Lingual Ticagrelor
- Sub Lingual Ticagrelor (Experimental)
  Interventions: Drug: Sub Lingual Ticagrelor

INTERVENTIONS:
Drug: Sub Lingual Ticagrelor — 180mg sub-lingual ticagrelor

SUMMARY:
Our goal is to examine sub lingual versus traditional oral administration of ticagrelor in ACS/non ST-elevation Myocardial Infarction (NSTEMI) patients on platelet reactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with ACS/NSTEMI
2. Informed, written consent

Exclusion Criteria:

1. Age < 18 years or Age > 90 years
2. Active bleeding; bleeding diathesis; coagulopathy
3. Increased risk of bradycardiac events
4. History of gastrointestinal or genitourinary bleeding <2 months
5. Major surgery in the last 6 weeks
6. History of intracranial bleeding or structural abnormalities
7. Suspected aortic dissection
8. Any other condition that may put the patient at risk or influence study results or investigator's opinion (severe hemodynamic instability, known malignancies or other comorbid conditions with life expectancy <1 year)
9. Administration in the week before the index event of clopidogrel, ticlopidine, prasugrel, ticagrelor, thrombolytics, bivalirudin, low-molecular weight heparin or fondaparinux.
10. Concomitant oral or IV therapy with strong CYP3A inhibitors or strong CYP3A inducers, CYP3A with narrow therapeutic windows
11. Known relevant hematological deviations: Hb <10 g/dl, PLT<100x10^9/l
12. Use of coumadin derivatives within the last 7 days
13. Chronic therapy with ticagrelor, prasugrel, clopidogrel or ticlopidine
14. Known severe liver disease, severe renal failure
15. Known allergy to the study medications
16. Pregnancy
17. Human immunodeficiency virus treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Residual platelet reactivity by Platelet Reactivity Units (PRU) VerifyNow 1 hour after ticagrelor LD | 1hour

SECONDARY OUTCOMES:
The percent of patients with a high residual platelet reactivity (PRU > 208) 1 hour, 4-6, 12 hours after ticagrelor LD. | 1, 4-6, 12 hours
Bleeding events: Major, minor, minimal bleeding (TIMI criteria) events. | 24 hours
Occurrence of dyspnea and/or symptomatic bradycardia. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical center, Ramat Gan, Israel

REFERENCES:
- [Derived] Asher E, Frydman S, Katz M, Regev E, Sabbag A, Mazin I, Abu-Much A, Kukuy A, Mazo A, Erez A, Berkovitch A, Narodistky M, Barbash I, Segev A, Beigel R, Matetzky S. Chewing versus Swallowing Ticagrelor to Accelerate Platelet Inhibition in Acute Coronary Syndrome - the CHEERS study. For The PLATIS (Platelets and Thrombosis in Sheba) Study Group. Thromb Haemost. 2017 Apr 3;117(4):727-733. doi: 10.1160/TH16-09-0728. Epub 2017 Feb 2. PMID 28150850